CLINICAL TRIAL: NCT02089139
Title: Intradiscal Injection of Gelified Ethanol for the Treatment of Discogenic Back Pain
Brief Title: Treatment of Discogenic Back Pain
Acronym: EGID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The French medicines agency did not allow the continuation of the study (no patient enrolled in this study)
Sponsor: University Hospital, Limoges (Other)
Collaborators: Gelscom SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I13009
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Discogenic Back Pain
Keywords: Back pain; Discogel
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DISCOGEL (Experimental): Percutaneous intradiscal injection of Discogel
  Interventions: Device: Discogel; Other: conventional treatment
- conventional treatment (Active Comparator): conventional treatment based on current guidelines regarding the management of discogenic low back pain, including but not limited to: medications (analgesics, NSAIDs, muscle relaxants), physical therapy, manual techniques, transcutaneous electrical nerve stimulation (TENS), blocks
  Interventions: Other: conventional treatment

INTERVENTIONS:
Device: Discogel — DiscoGel is a sterile viscous solution containing ethyl alcohol, cellulose derivative product and tungsten (radio-opaque element)
  Arms: DISCOGEL
Other: conventional treatment — Conventional treatment based on current guidelines regarding the management of discogenic low back pain, including but not limited to:
  * medications (analgesics, NSAIDs, muscle relaxants),
  * physical therapy,
  * manual techniques,
  * transcutaneous electrical nerve stimulation (TENS),
  * blocks

SUMMARY:
Discogenic low back pain is the most common form of chronic low back pain. Its diagnosis is mainly based on MR imaging, showing MODIC I or II changes in patients with concordant symptomatology. The treatment of discogenic low back pain is nevertheless difficult: intradiscal therapies (corticosteroids, methylene blue, radiofrequency) have a limited efficacy, and surgical procedures (arthrodesis or disc replacement) are a final recourse with notable risk of side-effects.

In this study, the efficacy of intradiscal injection of gelified ethanol (DiscoGel) in patients with disabling discogenic pain is assessed.

ELIGIBILITY:
Inclusion Criteria:

* MR imaging : MODIC 1or MODIC 2 changes limited to one single lumbar disc;
* X rays: normal disc height, no instability;
* Back pain for at least 3 months, without argument for another etiology;
* Mean pain on 5 days VAS ≥ 5

Exclusion Criteria:

* age <18 years or > 50 ; concomitant radicular pain ;
* psychiatric pathology that may modify the perception or the evolution of pain;
* MR imaging: multi-level discopathy, MODIC 3 changes;
* X ray: loss of disc height > 50%, segmental instability;
* previous history of lumbar surgery with or without instrumentation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Six months after the procedure.
  Mean pain intensity score on a Visual Analog Scale (VAS), six months after the procedure.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS), | one month, three months, six months and 1 year after the procedure
  Mean pain intensity score on Visual Analog Scale (VAS), one month, three months, six months and 1 year after the procedure ;
Oswestry Disability Index (ODI) | one month, three months, six months and 1 year after the procedure
  Oswestry Disability Index (ODI) one month, three months, six months and 1 year after the procedure ;
Euroqol score | month, three months, six months and 1 year after the procedure
  Assessment of the quality of life with Euroqol score (EQ-5D) one month, three months, six months and 1 year after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: CAIRE François, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- CHU Limoges, Limoges, France